CLINICAL TRIAL: NCT04750772
Title: Comparison of Positron Nuclide Labeled DOTA-FAPI PET and FDG PET Study in Colocrectal Cancer
Brief Title: Positron Nuclide Labeled DOTA-FAPI PET Study in Colocrectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xuejuan Wang,MD, Deputy Director of Nuclear Medicine, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: XW-YZ-FAPI-2019KT95
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Tumor, Solid; Positron-Emission Tomography; Colorectal Cancer
Keywords: Colorectal Cancer; Positron-Emission Tomography; FAPI
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-DOTA-FAPI04 (Experimental): Each subject receive a single intravenous injection of 18F-FDG and 68Ga-DOTA-FAPI04, and undergo PET/CT imaging within the specified time
  Interventions: Diagnostic Test: 18F-FDG and 68Ga-DOTA-FAPI04 PET/CT
- 18F-DOTA-FAPI04 (Experimental): Each subject receive a single intravenous injection of 18F-FDG and 18F-DOTA-FAPI04, and undergo PET/CT imaging within the specified time
  Interventions: Diagnostic Test: 18F-FDG and 18F-DOTA-FAPI04 PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG and 68Ga-DOTA-FAPI04 PET/CT — Each subject receive a single intravenous injection of 18F-FDG and 68Ga-DOTA-FAPI04, and undergo PET/CT imaging within the specified time
  Arms: 68Ga-DOTA-FAPI04
Diagnostic Test: 18F-FDG and 18F-DOTA-FAPI04 PET/CT — Each subject receive a single intravenous injection of 18F-FDG and 18F-DOTA-FAPI04, and undergo PET/CT imaging within the specified time
  Arms: 18F-DOTA-FAPI04

SUMMARY:
To evaluate the normal physiological distribution of positron nuclide labeled DOTA-FAPI PET/CT in human body and its diagnostic efficiency for colorectal cancers

DETAILED DESCRIPTION:
Participants first undergo an 18F-FDG PET/CT, followed by 68Ga-FAPI04 PET/CT in groups. The purpose of the study is to explore the possibility of superiority of FAPI in diagnosis of colorectal cancer (TNM staging) by the comparison of the two tracers uptake (the maximum of standardized uptake value, SUVmax). Histopathology and conventional imaging follow-up are served as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score 0-2
* patients with newly diagnosed or previously treated colorectal cancers
* patients who underwent paired 18F-FDG and 68Ga-FAPI PET/CT for tumor staging to decide the most proper treatment strategy
* patients who underwent paired 18F-FDG and 68Ga-FAPI PET/CT to detect tumor recurrence and metastases (repeat staging)
* expected survival ≥12 weeks
* blood routine, liver and kidney function meet the following criteria : blood routine: WBC≥4.0×109L or neutrophils ≥1.5×109L, PLT≥100×109/L, Hb≥90g/L;PT and APTT ULN 1.5 or less; Liver and kidney function: t-bil ≤1.5×ULT(upper limit of normal value), ALT/AST≤2.5ULN or ≤5×ULT(subjects with liver metastasis), ALP≤2.5ULN(ALP≤ 4.5ULN if there is bone metastasis or liver metastasis);BUN 1.5 x or less ULT, SCr 1.5 x or less ULT
* at least one measurable target lesion according to RECIST1.1
* women must use effective contraception during the study period and for 6 months after the end of the study (effective contraception means sterilization, hormone devices, condoms, contraceptives/pills, abstinence or vasectomy by a partner, etc.);Men should consent to subjects who must use contraception during the study period and for 6 months after the end of the study period
* able to understand and sign the informed consent voluntarily, with good compliance.

Exclusion Criteria:

* severe abnormalities of liver and kidney function;
* women preparing for pregnancy, pregnancy and lactation;
* cannot lie supine for half an hour;
* refuse to join the clinical researcher;
* suffering from claustrophobia or other mental illness;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
finial clinical staging（TNM） | 60-120days
  To explore the effect of FAPI PET/CT on staging of Colorectal cancer by comparing with FDG PET/CT

SECONDARY OUTCOMES:
SUVmax | 60-120days
  To compare the uptake （SUVmax）of two tracers （FAPI and FDG）in colorectal cancer (including the normal organs, primary tumors and metastases)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Yang, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loktev A, Lindner T, Burger EM, Altmann A, Giesel F, Kratochwil C, Debus J, Marme F, Jager D, Mier W, Haberkorn U. Development of Fibroblast Activation Protein-Targeted Radiotracers with Improved Tumor Retention. J Nucl Med. 2019 Oct;60(10):1421-1429. doi: 10.2967/jnumed.118.224469. Epub 2019 Mar 8. PMID 30850501
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Result] Dekker E, Tanis PJ, Vleugels JLA, Kasi PM, Wallace MB. Colorectal cancer. Lancet. 2019 Oct 19;394(10207):1467-1480. doi: 10.1016/S0140-6736(19)32319-0. PMID 31631858
- [Result] Chakedis J, Schmidt CR. Surgical Treatment of Metastatic Colorectal Cancer. Surg Oncol Clin N Am. 2018 Apr;27(2):377-399. doi: 10.1016/j.soc.2017.11.010. Epub 2017 Dec 15. PMID 29496096
- [Result] Kantorova I, Lipska L, Belohlavek O, Visokai V, Trubac M, Schneiderova M. Routine (18)F-FDG PET preoperative staging of colorectal cancer: comparison with conventional staging and its impact on treatment decision making. J Nucl Med. 2003 Nov;44(11):1784-8. PMID 14602860
- [Result] Petersen RK, Hess S, Alavi A, Hoilund-Carlsen PF. Clinical impact of FDG-PET/CT on colorectal cancer staging and treatment strategy. Am J Nucl Med Mol Imaging. 2014 Aug 15;4(5):471-82. eCollection 2014. PMID 25143865
- [Result] Berger KL, Nicholson SA, Dehdashti F, Siegel BA. FDG PET evaluation of mucinous neoplasms: correlation of FDG uptake with histopathologic features. AJR Am J Roentgenol. 2000 Apr;174(4):1005-8. doi: 10.2214/ajr.174.4.1741005. PMID 10749239
- [Result] Borello A, Russolillo N, Lo Tesoriere R, Langella S, Guerra M, Ferrero A. Diagnostic performance of the FDG-PET/CT in patients with resected mucinous colorectal liver metastases. Surgeon. 2021 Oct;19(5):e140-e145. doi: 10.1016/j.surge.2020.09.004. Epub 2020 Oct 23. PMID 34581274
- [Result] Lindner T, Loktev A, Altmann A, Giesel F, Kratochwil C, Debus J, Jager D, Mier W, Haberkorn U. Development of Quinoline-Based Theranostic Ligands for the Targeting of Fibroblast Activation Protein. J Nucl Med. 2018 Sep;59(9):1415-1422. doi: 10.2967/jnumed.118.210443. Epub 2018 Apr 6. PMID 29626119
- [Result] Chen H, Pang Y, Wu J, Zhao L, Hao B, Wu J, Wei J, Wu S, Zhao L, Luo Z, Lin X, Xie C, Sun L, Lin Q, Wu H. Comparison of [68Ga]Ga-DOTA-FAPI-04 and [18F] FDG PET/CT for the diagnosis of primary and metastatic lesions in patients with various types of cancer. Eur J Nucl Med Mol Imaging. 2020 Jul;47(8):1820-1832. doi: 10.1007/s00259-020-04769-z. Epub 2020 Mar 28. PMID 32222810